CLINICAL TRIAL: NCT07259954
Title: Prediabetes Among Young Adults and Its Relation to Metabolic Parameters in Persons Attending Assuit University Hospital
Brief Title: Prediabetes and Metabolic Parameters Among Young Adults at Assiut University Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba Gamal Ali Mohamed, Internal medicine ,assuit university hospital, Assiut University
Other Study IDs: AUH-MED-PREDIAB-2025
Record Dates: First submitted 2025-09-14; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: PreDiabetes
Keywords: Predabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group A impaired glucose tolerance_Group B - Impaired Fasting Glucose Group C - Impaired HbA1c
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Participants will be classified into groups based on impaired fasting glucose, impaired post-prandial glucose, or impaired HbA1c according to ADA criteria

SUMMARY:
Prediabetes is a major public health problem that increases the risk of developing type 2 diabetes mellitus and cardiovascular complications. Young adults represent an important age group in which early detection and intervention may prevent progression of the disease. The present study aims to identify factors associated with prediabetes and metabolic complications, and classify individuals based on clinical and biochemical profiles according to insulin resistance, dyslipidemia and fatty liver. This is an observational, cross-sectional study that will be conducted at Assiut University Hospital. Data will be collected through clinical examination, laboratory investigations, and assessment of metabolic profiles.

ELIGIBILITY:
Inclusion Criteria:

* adults diagnosed with prediabetes

Exclusion Criteria:

* previous diagnosis of overt diabetes
* other causes of CKD (e.g. urinary tract infection)
* other causes of liver disease (e.g. HBV infection),
* use of medications that alter glucose or lipid metabolism (e.g. corticosteroids),
* current pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of young adults aged 18-40 years attending outpatient clinics at Assiut University Hospital. Participants will be screened for prediabetes using fasting plasma glucose, 2-hour postprandial glucose, and HbA1c tests. Only individuals diagnosed with prediabetes according to ADA criteria (impaired fasting glucose, impaired glucose tolerance, or elevated HbA1c) will be included
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between prediabetes subtypes and metabolic syndrome | At baseline (cross-sectional assessment during enrollment).
  Primary Outcome
  Title:
  Correlation between prediabetes phenotypes and metabolic syndrome
  Outcome Measure:
  Prevalence (%) of metabolic syndrome within each prediabetes phenotype (IFG, IGT, combined IFG/IGT, elevated HbA1c).
  Description:
  Metabolic syndrome will be assessed at baseline according to the IDF definition. Participants will be classified into prediabetes phenotypes, and the proportion of individuals meeting metabolic syndrome criteria within each phenotype will be recorded.
  Time Frame:
  Baseline
  Unit of Measure:
  Percentage (%)

SECONDARY OUTCOMES:
Factors affecting the correlation between prediabetes phenotypes and metabolic abnormalities (age, gender, family history, body physique, waist circumference and physical activity. | At baseline (cross-sectional assessment during enrollment)
  Secondary Outcome 1 Title: Age Description: Participant age in years. Unit of Measure: Years Time Frame: Baseline Secondary Outcome 2 Title: Sex Description: Participant sex as recorded at baseline. Unit of Measure: Categorical Time Frame: Baseline Secondary Outcome 3 Title: Family history of diabetes Description: Presence of family history of diabetes in first-degree relatives. Unit of Measure: Yes/No Time Frame: Baseline Secondary Outcome 4 Title: Weight Description: Body weight measured using a calibrated scale. Unit of Measure: Kilograms Time Frame: Baseline Secondary Outcome 5 Title: Height Description: Participant height measured using a stadiometer. Unit of Measure: Centimeters Time Frame: Baseline Secondary Outcome 6 Title: Body Mass Index (BMI) Description: BMI calculated as weight (kg) divided by height squared (m²). Unit of Measure: kg/m² Time Frame: Baseline Secondary Outcome 7 Title: Waist circumference Description: Waist circumference measured using a non-stretchab

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] http://doi.org/10.1007/s00125-013-2902-4
- [Background] http://doi.org/10.1136/bmj.g4485
- [Background] http://doi.org/10.1007/s00125-009-1443-3
- [Background] http://doi.org/10.2337/dc08-1264
- [Background] http://doi.org/10.1016/j.diabres.2007.05.004
- [Background] http://doi.org/10.2337/diabetes.52.6.1475
- [Background] http://doi.org/10.1136/bmj.i5953
- [Background] http://doi.org/10.1056/NEJMoa012512
- [Background] http://doi.org/10.1016/S0140-6736(12)60525-X
- [Background] http://doi.org/10.2337/dc10-0679
- [Background] http://doi.org/10.2337/diacare.2951130
- [Background] http://doi.org/10.2337/dc07-9920
- [Background] http://doi.org/10.1016/S0140-6736(12)60283-9
- [Background] International Diabetes Federation. IDF Diabetes Atlas. 10th ed. Brussels: IDF; 2021. http://www.diabetesatlas.org
- See also: Related Info — http://www.diabetesatlas.org
- See also: Related Info — http://doi.org/10.1016/S0140-6736(12)60283-9
- See also: Related Info — http://doi.org/10.1007/s00125-009-1443-3